CLINICAL TRIAL: NCT02469428
Title: Epigenetic Effect Modifications With Ozone Exposure on Healthy Volunteers
Acronym: Geminoz
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Environmental Protection Agency (EPA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, David Diaz-Sanchez, Principal Investigator, Environmental Protection Agency (EPA)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 13-3697
Record Dates: First submitted 2015-06-05; First posted 2015-06-11 (Estimated); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Exposure to Environmental Pollution, Non-occupational
Keywords: Controlled human exposure study; Ozone; Inflammation
MeSH Terms: conditions — Inflammation | interventions — Environment, Controlled; Ozone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clean air (Sham Comparator): Exposure to clean air will be conducted in an exposure chamber at the EPA Human Studies Facility on the UNC campus.
  Interventions: Other: Clean air
- Ozone (Experimental): Exposure to ozone will be conducted in an exposure chamber at the EPA Human Studies Facility on the UNC campus.
  Interventions: Other: Ozone

INTERVENTIONS:
Other: Clean air — Each subject will be exposed to clean air for 2 hours. Subjects will exercise on a bike. Each exercise session will consist of a 15 minute exercise interval at a level of up to 20 L/min/m2 BSA followed by a 15 minute rest period, repeated 4 times.
  Arms: Clean air
Other: Ozone — Each subject will be exposed to 0.3 ppb ozone for 2 hours. Subjects will exercise on a bike. Each exercise session will consist of a 15 minute exercise interval at a level of up to 20 L/min/m2 BSA followed by a 15 minute rest period, repeated 4 times.
  Arms: Ozone

SUMMARY:
The purpose of this protocol is to assess whether epigenetic factors in healthy individuals make a person more or less responsive to lung inflammation following ozone exposures.

DETAILED DESCRIPTION:
Controlled human exposure studies to ozone have reported decreases in lung function (Devlin et al. 2012; Kim et al. 2011) and increased inflammation (Kim et al. 2011; Koren et al. 1991; Liu et al. 2009; Romieu et al. 2008). However, the range of response to ozone in healthy young volunteers is an order of magnitude, and if individuals are exposed to ozone some months later they retain their hierarchy on the response curve, suggesting that long-lived factors are responsible. Several studies have demonstrated that polymorphisms in oxidative stress genes such as GSTM1 or NQO1 may be associated with responsiveness to air pollutants (Bergamaschi et al. 2001; Corradi et al. 2002). However, within the past decade, many researchers have started exploring the epigenome as a possible link between exposures to environmental toxicants and disease. Epigenetics refers to non-genetic mechanisms influencing gene expression and phenotype (Cortessis et al. 2012). Commonly studied epigenetic changes include DNA methylation, histone modification, and non-coding RNA expression (i.e. micro-RNA). Recently, work conducted at the Harvard School of Public Health looked at DNA methylation as an effect modifier to air pollution-induced adverse health effects (Bind et al. 2012). This group, using a cohort representing previous war veterans from the VA Normative Aging Study, observed stronger effects in cardiovascular disease-related blood biomarkers with DNA methylation status, both globally and within candidate genes. Additionally, Salam et al. found that fractional exhaled nitric oxide, a marker of lung inflammation, was interrelated with short-term PM 2.5 concentration as well as NOS2 epigenetic and genetic variations in children (2012). Thus, these studies suggest epigenetic changes could impact susceptibility to pollutants. Additionally, acute epigenetic changes, which are potential pathways of air pollution-induced health effects, have been associated with the inhalation of particulate matter and ambient gaseous pollutants (Baccarelli et al. 2009; Bellavia et al. 2013; Bollati et al. 2010; De Prins et al. 2013; Madrigano et al. 2011; Tarantini et al. 2009). Therefore, it is possible that an individual's epigenetic profile could make them more or less responsive to ozone, and that ozone exposure itself could cause acute changes in the epigenome which could in turn affect ozone-responsiveness.

Previous studies that have looked at epigenetic changes associated with air pollutants have difficultly disentangling the role of genetic and epigenetic factors. One way to do this is to study identical (MZ) twins. MZ twins arise when two or more daughter cells split from a single zygote during embryonic development, forming two individuals with identical genetic sequences (Fraga et al. 2005) but dissimilar epigenomes (Li et al. 2013; Szyf 2007). A number of diseases in which MZ twins are discordant, such as bipolar and schizophrenia disorders (Bonsch et al. 2012; Dempster et al. 2011), asthma (Runyon et al. 2012), autism spectrum disorder (Wong et al. 2013), and breast cancer (Heyn et al. 2013), implicate epigenetic variability as the cause. Therefore, as discordance for disease status has already been linked with epigenetic changes, this adds further plausibility to the notion that epigenetics could be responsible for the susceptibility of some subjects to ozone exposures while others seem non-responsive. By using MZ twins as one target population for this study, variability due only to epigenetics, without the influence of genetics, can be fully explored.

For this study, the investigators will measure changes in pulmonary inflammation after a controlled exposure in healthy subjects and healthy twin pairs to clean air and ozone. This endpoint was chosen because previous work has shown that the epithelial cells lining the airways are the first target of ozone and respond by making pro-inflammatory cytokines such as IL-6 and IL-8. Epigenetic changes are dependent on tissue type, and airway epithelial cells can be obtained by brush biopsies during bronchoscopy and assayed for epigenetic changes. The investigators will determine whether differences in baseline epigenetic profiles between subjects are associated with responsiveness to ozone and whether ozone exposure itself causes acute changes in a subject's epigenome.

ELIGIBILITY:
Inclusion Criteria:

1. Normal baseline 12-lead resting EKG.
2. Normal lung function, defined by NHANES III as:

   * FVC of > 80 %.
   * FEV1 of > 80 %.
   * FEV1/FVC ratio of > 80 %.
3. Oxygen saturation of > 96 %.
4. Ability to complete the exposure exercise regimen without reaching 80% of predicted maximal heart rate.

Exclusion Criteria:

1. A history of acute and/or chronic illnesses such as diabetes, rheumatological diseases, immunodeficiency state, neurological disease, renal disease, liver disease, endocrinological disease, malignancy, cardiovascular disease, chronic respiratory diseases, and lung cancer.
2. Asthma or a history of asthma.
3. A Framingham risk score ≥10.
4. Women who are pregnant, attempting to become pregnant, or breastfeeding.
5. An allergy to any medications which may be used or prescribed in the course of this study.
6. Cannot refrain from taking vitamins C or E (or multivitamins which contain Vitamins C or E) for 7 days prior to all visits.
7. Cannot refrain from taking supplements for 7 days prior to all visits that contain homeopathic/naturopathic medicines or medications which may impact the results of the ozone challenge or interfere with any other medications potentially used in the study. Medications not specifically mentioned here may be reviewed by the investigators and medical staff prior to inclusion in the study.
8. Untreated hypertension (≥ 150 systolic or ≥ 90 diastolic blood pressure).
9. Dementia.
10. Unspecified illnesses, which in the judgment of the investigator or medical staff might increase the risk associated ozone inhalation challenge or exercise.
11. A history of skin allergies to adhesives used in securing EKG electrodes.
12. Do not understand or speak English.
13. Chronic and continuous allergic rhinitis.
14. Unable to perform the moderate exercise required for the study.
15. Those that are unwilling or unable to refrain from the following medications for the week prior to each exposure: anti-inflammatory agents such as ibuprofen, naproxen, or aspirin.
16. Those currently taking or have taken anti-coagulant medication in the week prior to each exposure.
17. Currently smoker or has a smoked within the last 2 years, or if you have a smoking history > 1 pack-years or are living with a smoker that smokes inside the house.
18. A history of fainting in response to blood being drawn or other medical procedures.
19. Unwilling or unable to stay for a suitable observation period after the procedure at the discretion of the physician involved, and not ride a bicycle or motorcycle home.
20. You are unwilling or unable to refrain from strenuous exercise for 24 hours prior to and after all visits, consuming caffeine for 12 hours prior to all study visits, using of antihistamines for one week prior to exposures, and drinking alcohol 24 hours before all visits.

Temporary exclusions:

1. Viral upper respiratory tract infection or any acute infection within 6 weeks of bronchoscopy.
2. Current exacerbation of allergic rhinitis and or use of antihistamines during one week prior to exposure.
3. Recent or recurring exposure to pollutants or irritants.

Exclusion criteria for bronchoscopy:

1. Any food or fluids after midnight prior to bronchoscopy.
2. FEV1 decrement of >10% from baseline on AM of bronchoscopy.
3. Use of aspirin ≥ 81 mg daily, or other nonsteroidal anti-inflammatory drugs within one week of bronchoscopy.
4. You are unwilling or unable to take nothing by mouth after midnight the night before bronchoscopy.
5. You are unwilling or unable to stay in the local Raleigh/Durham/Chapel Hill area for 24 hours after the procedure.

Use of other medications will be evaluated on a case-by-case basis. There is the potential that an individual's current medication use will preclude them from participating in the study at the current time, but they may be reassessed and potentially rescheduled for participation at a later time.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2013-12; Primary Completion 2017-07 (Actual); Study Completion 2018-11-05 (Actual)

PRIMARY OUTCOMES:
Pulmonary inflammation | pre-exposure to 18 hrs post exposure
  18 hrs following exposures the subjects will undergo a research bronchoscopy where lavage fluid and epithelial cells via brush biopsy will be collected. Protein content will be assessed in lavage fluid. Changes in inflammatory genes will be measured in epithelial cells. DNA will be extracted from epithelial cells and DNA methylation arrays will be run.

SECONDARY OUTCOMES:
Changes in heart rate variability | pre-exposure to 18 hrs post-exposure
  10 minute electrocardiogram recording (measured by Holter ECG) in which the subject has been resting for 20 minutes prior. Collected on a Mortara H12+ 12-lead ECG recorder. The digitally recorded ECGs are sampled at 180 Hz.
Forced expiratory volume in 1 second (FEV1) | pre-exposure to 18 hrs post-exposure
  FEV1 is determined by spirometry performed on a dry seal spirometer interfaced to a computer.
Forced vital capacity (FVC) | pre-exposure to 18 hrs post-exposure
  FVC is determined by spirometry performed on a dry seal spirometer interfaced to a computer.
Index of clotting/coagulation factors | pre-exposure to 18 hrs post-exposure
  Index of clotting/coagulation factors are the mean percent changes in a variety of clotting/coagulation factors (d-dimer, PA-1, tPA, vWillebrand factor, plasminogen) in the blood.
Index of inflammatory factors from blood | pre-exposure to 18 hrs post-exposure
  Index of inflammatory factors are the mean percent changes in a variety of systemic inflammatory factors (IL-6, IL-8, TNF-a, IL-1b, CRP) in the blood.

CONTACTS AND LOCATIONS:
Overall Officials: David Diaz-Sanchez, PhD, Principal Investigator — Environmental Protection Agency (EPA)
Locations (1):
- EPA Human Studies Facility, Chapel Hill, North Carolina, United States

REFERENCES:
- [Background] Baccarelli A, Wright RO, Bollati V, Tarantini L, Litonjua AA, Suh HH, Zanobetti A, Sparrow D, Vokonas PS, Schwartz J. Rapid DNA methylation changes after exposure to traffic particles. Am J Respir Crit Care Med. 2009 Apr 1;179(7):572-8. doi: 10.1164/rccm.200807-1097OC. Epub 2009 Jan 8. PMID 19136372
- [Background] Bellavia A, Urch B, Speck M, Brook RD, Scott JA, Albetti B, Behbod B, North M, Valeri L, Bertazzi PA, Silverman F, Gold D, Baccarelli AA. DNA hypomethylation, ambient particulate matter, and increased blood pressure: findings from controlled human exposure experiments. J Am Heart Assoc. 2013 Jun 19;2(3):e000212. doi: 10.1161/JAHA.113.000212. PMID 23782920
- [Background] Bergamaschi E, De Palma G, Mozzoni P, Vanni S, Vettori MV, Broeckaert F, Bernard A, Mutti A. Polymorphism of quinone-metabolizing enzymes and susceptibility to ozone-induced acute effects. Am J Respir Crit Care Med. 2001 May;163(6):1426-31. doi: 10.1164/ajrccm.163.6.2006056. PMID 11371413
- [Background] Bind MA, Baccarelli A, Zanobetti A, Tarantini L, Suh H, Vokonas P, Schwartz J. Air pollution and markers of coagulation, inflammation, and endothelial function: associations and epigene-environment interactions in an elderly cohort. Epidemiology. 2012 Mar;23(2):332-40. doi: 10.1097/EDE.0b013e31824523f0. PMID 22237295
- [Background] Bollati V, Marinelli B, Apostoli P, Bonzini M, Nordio F, Hoxha M, Pegoraro V, Motta V, Tarantini L, Cantone L, Schwartz J, Bertazzi PA, Baccarelli A. Exposure to metal-rich particulate matter modifies the expression of candidate microRNAs in peripheral blood leukocytes. Environ Health Perspect. 2010 Jun;118(6):763-8. doi: 10.1289/ehp.0901300. Epub 2010 Jan 8. PMID 20061215
- [Background] Bonsch D, Wunschel M, Lenz B, Janssen G, Weisbrod M, Sauer H. Methylation matters? Decreased methylation status of genomic DNA in the blood of schizophrenic twins. Psychiatry Res. 2012 Aug 15;198(3):533-7. doi: 10.1016/j.psychres.2011.09.004. Epub 2012 Oct 25. PMID 23102571
- [Background] Corradi M, Alinovi R, Goldoni M, Vettori M, Folesani G, Mozzoni P, Cavazzini S, Bergamaschi E, Rossi L, Mutti A. Biomarkers of oxidative stress after controlled human exposure to ozone. Toxicol Lett. 2002 Aug 5;134(1-3):219-25. doi: 10.1016/s0378-4274(02)00169-8. PMID 12191881
- [Background] Cortessis VK, Thomas DC, Levine AJ, Breton CV, Mack TM, Siegmund KD, Haile RW, Laird PW. Environmental epigenetics: prospects for studying epigenetic mediation of exposure-response relationships. Hum Genet. 2012 Oct;131(10):1565-89. doi: 10.1007/s00439-012-1189-8. Epub 2012 Jun 28. PMID 22740325
- [Background] De Prins S, Koppen G, Jacobs G, Dons E, Van de Mieroop E, Nelen V, Fierens F, Int Panis L, De Boever P, Cox B, Nawrot TS, Schoeters G. Influence of ambient air pollution on global DNA methylation in healthy adults: a seasonal follow-up. Environ Int. 2013 Sep;59:418-24. doi: 10.1016/j.envint.2013.07.007. Epub 2013 Aug 3. PMID 23917442
- [Background] Dempster EL, Pidsley R, Schalkwyk LC, Owens S, Georgiades A, Kane F, Kalidindi S, Picchioni M, Kravariti E, Toulopoulou T, Murray RM, Mill J. Disease-associated epigenetic changes in monozygotic twins discordant for schizophrenia and bipolar disorder. Hum Mol Genet. 2011 Dec 15;20(24):4786-96. doi: 10.1093/hmg/ddr416. Epub 2011 Sep 9. PMID 21908516
- [Background] Devlin RB, Duncan KE, Jardim M, Schmitt MT, Rappold AG, Diaz-Sanchez D. Controlled exposure of healthy young volunteers to ozone causes cardiovascular effects. Circulation. 2012 Jul 3;126(1):104-11. doi: 10.1161/CIRCULATIONAHA.112.094359. Epub 2012 Jun 25. PMID 22732313
- [Background] Fraga MF, Ballestar E, Paz MF, Ropero S, Setien F, Ballestar ML, Heine-Suner D, Cigudosa JC, Urioste M, Benitez J, Boix-Chornet M, Sanchez-Aguilera A, Ling C, Carlsson E, Poulsen P, Vaag A, Stephan Z, Spector TD, Wu YZ, Plass C, Esteller M. Epigenetic differences arise during the lifetime of monozygotic twins. Proc Natl Acad Sci U S A. 2005 Jul 26;102(30):10604-9. doi: 10.1073/pnas.0500398102. Epub 2005 Jul 11. PMID 16009939
- [Background] Heyn H, Carmona FJ, Gomez A, Ferreira HJ, Bell JT, Sayols S, Ward K, Stefansson OA, Moran S, Sandoval J, Eyfjord JE, Spector TD, Esteller M. DNA methylation profiling in breast cancer discordant identical twins identifies DOK7 as novel epigenetic biomarker. Carcinogenesis. 2013 Jan;34(1):102-8. doi: 10.1093/carcin/bgs321. Epub 2012 Oct 10. PMID 23054610
- [Background] Kim CS, Alexis NE, Rappold AG, Kehrl H, Hazucha MJ, Lay JC, Schmitt MT, Case M, Devlin RB, Peden DB, Diaz-Sanchez D. Lung function and inflammatory responses in healthy young adults exposed to 0.06 ppm ozone for 6.6 hours. Am J Respir Crit Care Med. 2011 May 1;183(9):1215-21. doi: 10.1164/rccm.201011-1813OC. Epub 2011 Jan 7. PMID 21216881
- [Background] Koren HS, Devlin RB, Becker S, Perez R, McDonnell WF. Time-dependent changes of markers associated with inflammation in the lungs of humans exposed to ambient levels of ozone. Toxicol Pathol. 1991;19(4 Pt 1):406-11. doi: 10.1177/0192623391019004-109. PMID 1813985
- [Background] Li C, Zhao S, Zhang N, Zhang S, Hou Y. Differences of DNA methylation profiles between monozygotic twins' blood samples. Mol Biol Rep. 2013 Sep;40(9):5275-80. doi: 10.1007/s11033-013-2627-y. Epub 2013 May 7. PMID 23649773
- [Background] Liu L, Poon R, Chen L, Frescura AM, Montuschi P, Ciabattoni G, Wheeler A, Dales R. Acute effects of air pollution on pulmonary function, airway inflammation, and oxidative stress in asthmatic children. Environ Health Perspect. 2009 Apr;117(4):668-74. doi: 10.1289/ehp11813. Epub 2008 Nov 28. PMID 19440509
- [Background] Madrigano J, Baccarelli A, Mittleman MA, Wright RO, Sparrow D, Vokonas PS, Tarantini L, Schwartz J. Prolonged exposure to particulate pollution, genes associated with glutathione pathways, and DNA methylation in a cohort of older men. Environ Health Perspect. 2011 Jul;119(7):977-82. doi: 10.1289/ehp.1002773. Epub 2011 Mar 8. PMID 21385671
- [Background] Romieu I, Barraza-Villarreal A, Escamilla-Nunez C, Almstrand AC, Diaz-Sanchez D, Sly PD, Olin AC. Exhaled breath malondialdehyde as a marker of effect of exposure to air pollution in children with asthma. J Allergy Clin Immunol. 2008 Apr;121(4):903-9.e6. doi: 10.1016/j.jaci.2007.12.004. Epub 2008 Jan 30. PMID 18234317
- [Background] Runyon RS, Cachola LM, Rajeshuni N, Hunter T, Garcia M, Ahn R, Lurmann F, Krasnow R, Jack LM, Miller RL, Swan GE, Kohli A, Jacobson AC, Nadeau KC. Asthma discordance in twins is linked to epigenetic modifications of T cells. PLoS One. 2012;7(11):e48796. doi: 10.1371/journal.pone.0048796. Epub 2012 Nov 30. PMID 23226205
- [Background] Salam MT, Byun HM, Lurmann F, Breton CV, Wang X, Eckel SP, Gilliland FD. Genetic and epigenetic variations in inducible nitric oxide synthase promoter, particulate pollution, and exhaled nitric oxide levels in children. J Allergy Clin Immunol. 2012 Jan;129(1):232-9.e1-7. doi: 10.1016/j.jaci.2011.09.037. Epub 2011 Nov 4. PMID 22055874
- [Background] Szyf M. The dynamic epigenome and its implications in toxicology. Toxicol Sci. 2007 Nov;100(1):7-23. doi: 10.1093/toxsci/kfm177. Epub 2007 Aug 3. PMID 17675334
- [Background] Tarantini L, Bonzini M, Apostoli P, Pegoraro V, Bollati V, Marinelli B, Cantone L, Rizzo G, Hou L, Schwartz J, Bertazzi PA, Baccarelli A. Effects of particulate matter on genomic DNA methylation content and iNOS promoter methylation. Environ Health Perspect. 2009 Feb;117(2):217-22. doi: 10.1289/ehp.11898. Epub 2008 Sep 26. PMID 19270791
- [Background] Wong CC, Meaburn EL, Ronald A, Price TS, Jeffries AR, Schalkwyk LC, Plomin R, Mill J. Methylomic analysis of monozygotic twins discordant for autism spectrum disorder and related behavioural traits. Mol Psychiatry. 2014 Apr;19(4):495-503. doi: 10.1038/mp.2013.41. Epub 2013 Apr 23. PMID 23608919